CLINICAL TRIAL: NCT02376504
Title: Modifying the Workplace to Decrease Sedentary Behavior and Improve Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Dinesh John, Assistant Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21OH010564-01 (NIH)
Record Dates: First submitted 2015-02-20; First posted 2015-03-03 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Workplace Inactivity; Total Worker Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treadmill workstation (Experimental): Participants will be provided with a treadmill workstation to be more active at the workplace Active Workplace
  Interventions: Behavioral: Active workplace
- Sit-to-Stand workstation (Experimental): Participants will be provided with a sit-to-stand workstation to be decrease sitting time at the workplace Active Workplace
  Interventions: Behavioral: Active workplace
- Control (No Intervention): Participants will be asked to engage in three 10 min walking bouts each work day

INTERVENTIONS:
Behavioral: Active workplace — This is a 12-month, cluster-randomized trial with an intent-to-treat design to determine the effects of using treadmill and sit-to-stand workstations at the workplace on health variables in overweight office workers (N=66) with seated desk jobs and (2) to compare the efficacies of treadmill and sit-to-stand workstations in decreasing workplace sedentary behavior. The intervention will examine the effects of using these workstations on weight, cardiovascular and metabolic health variables , musculoskeletal discomfort, psychological affect and job stress. The study will also measure change in time spent sitting, standing and walking will be measured using wearable non-invasive acceleration sensors.
  Arms: Sit-to-Stand workstation; Treadmill workstation

SUMMARY:
The primary objective of this project is to determine the effects of decreasing sedentary behavior at work by at least 3hrs/day using treadmill (walking and standing) and sit-to-stand (standing only) workstations on the health of overweight office workers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than 25 kg.m-2
* Does not engage in any structured physical activity lasting at least 30 mins for more than 2 days/week
* Employed in a full-time sedentary desk job.
* No major orthopedic limitations or medical conditions that prevents walking or standing at a treadmill work sit-stand workstation.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 3, 6, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh John, PhD, Principal Investigator — Northeastern University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Arguello D, Cloutier G, Thorndike AN, Castaneda Sceppa C, Griffith J, John D. Impact of Sit-to-Stand and Treadmill Desks on Patterns of Daily Waking Physical Behaviors Among Overweight and Obese Seated Office Workers: Cluster Randomized Controlled Trial. J Med Internet Res. 2023 May 16;25:e43018. doi: 10.2196/43018. PMID 37191995
- [Derived] Arguello D, Thorndike AN, Cloutier G, Morton A, Castaneda-Sceppa C, John D. Effects of an "Active-Workstation" Cluster RCT on Daily Waking Physical Behaviors. Med Sci Sports Exerc. 2021 Jul 1;53(7):1434-1445. doi: 10.1249/MSS.0000000000002594. PMID 33449603